CLINICAL TRIAL: NCT00592839
Title: A Phase 4, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Effects of SCE-B on Nocturnal Vasomotor Symptoms in Postmenopausal Women
Brief Title: Study to Evaluate the Effects of Synthetic Conjugated Estrogens, B (SCE-B) on Nocturnal Vasomotor Symptoms in Postmenopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duramed Research (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DR-ENJ-401
Record Dates: First submitted 2007-12-20; First posted 2008-01-14 (Estimated); Results first posted 2010-03-17 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Nocturnal Vasomotor Symptoms
Keywords: Nocturnal vasomotor symptoms in postmenopausal women
MeSH Terms: interventions — estrogens, conjugated synthetic B

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): 0.3 mg SCE-B Daily
  Interventions: Drug: SCE-B; Drug: Placebo
- 2 (Experimental): 0.625 mg SCE-B Daily
  Interventions: Drug: SCE-B; Drug: Placebo
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SCE-B — 0.3 mg or 0.625 mg SCE-B tablets daily plus matching placebo
  Other Names: Synthetic Conjugated Estrogens, B; Enjuvia
  Arms: 1; 2
Drug: Placebo — Matching placebo for 0.3 mg and 0.625 mg tablets

SUMMARY:
This is a multi-center study to evaluate the effects of SCE-B on nocturnal vasomotor symptoms. Study duration will be approximately 16 weeks; this includes a 4-week screening period and approximately 5 scheduled clinic visits. Participants will receive one of two strengths of SCE-B tablets plus matching placebo or placebo only, and will have a physical and gynecological exams that may include transvaginal ultrasound, endometrial biopsy and a pap smear. Participants will be asked to wear a monitoring device for a portion of the study and be asked to complete a daily dairy.

ELIGIBILITY:
Inclusion Criteria:

* Naturally or surgically menopausal
* Minimum 7 daily or 50 weekly moderate-to-severe hot flashes

Exclusion Criteria:

* Any contraindication to hormone therapy

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2007-12; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Protocol Chair, Study Chair — Duramed Research, Inc.
Locations (17):
- United States (17):
  - Duramed Investigational Site, Anaheim, California
  - Duramed Investigational Site, Sacramento, California
  - Duramed Investigational Site, San Diego, California
  - Duramed Investigational Site, Clearwater, Florida
  - Duramed Investigational Site, West Palm Beach, Florida
  - Duramed Investigational Site, Lexington, Kentucky
  - Duramed Investigational Site, Louisville, Kentucky
  - Duramed Investigational Site, Lincoln, Nebraska
  - Duramed Investigational Site, Moorestown, New Jersey
  - Duramed Investigational Site, Albuquerque, New Mexico
  - Duramed Investigational Site, Winston-Salem, North Carolina
  - Duramed Investigational Site, Cleveland, Ohio
  - Duramed Investigational Site, Mayfield Heights, Ohio
  - Duramed Investigational Site, Medford, Oregon
  - Duramed Investigational Site, Pittsburgh, Pennsylvania
  - Duramed Investigational Site, Columbia, South Carolina
  - Duramed Investigational Site, San Antonio, Texas

REFERENCES:
- [Derived] Liu JH, Reape KZ, Hait HI. Synthetic conjugated estrogens-B and postmenopausal nocturnal vasomotor symptoms: a randomized controlled trial. Obstet Gynecol. 2012 Jan;119(1):78-84. doi: 10.1097/AOG.0b013e31823c0145. PMID 22183214

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.3 mg SCE-B Daily: SCE-B tablet 0.3 mg/day orally
- 0.625 mg SCE-B Daily: SCE-B tablet 0.625 mg/day orally
- Placebo Daily: Placebo tablet daily orally
Period: Overall Study
Arm/Group | 0.3 mg SCE-B Daily | 0.625 mg SCE-B Daily | Placebo Daily
Started | 53 | 52 | 52
Completed | 51 | 48 | 46
Not Completed | 2 | 4 | 6
Not completed — Withdrawal by Subject | 1 | 1 | 3
Not completed — Protocol Violation | 1 | 1 | 2
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.3 mg SCE-B Daily | 0.625 mg SCE-B Daily | Placebo Daily | Total
Number analyzed (Participants) | 53 | 52 | 52 | 157
Age, Customized [Number; unit: participants]
  Between 30 and 65 years | 53 | 52 | 52 | 157
Age Continuous [Mean (Standard Deviation); unit: years] | 53.9 (6.00) | 54.6 (5.38) | 53.8 (6.27) | 54.1 (5.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 52 | 52 | 157
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 53 | 52 | 52 | 157

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Average Frequency of Awakenings Due to Sleep-time Hot Flashes
Description: Change= Week 12 weekly average awakening score - Baseline weekly average awakening score for the intent-to-treat cohort
Time Frame: Baseline to End of Treatment (Week 12)
Population: Participants analyzed consisted of subjects from the intent-to-treat (ITT) cohort, [all subjects who were exposed to investigational product therapy,provided baseline "sleep time" hot flash information and "sleep time" hot flash data for at least one post-baseline visit]. Not all study subjects completed all data elements in their study diaries.
Measure: Least Squares Mean (Standard Error); unit: Awakenings
Arm/Group | 0.3 mg SCE-B Daily | 0.625 mg SCE-B Daily | Placebo Daily
Number analyzed (Participants) | 52 | 48 | 51
Awakenings | -19.54 (1.195) | -20.55 (1.286) | -15.99 (1.234)

2. Secondary Outcome: Mean Change in Individual Sleep Parameters on a Three-point Scale
Description: Change= Week 12 weekly average sleep quality score - Baseline weekly average sleep quality score for the intent-to-treat cohort. The sleep quality was derived from the subject self-assessment of sleep quality graded on a three-point scale (3=excellent, 2=good, 1=poor sleep quality)
Time Frame: Baseline to End of Treatment (Week 12)
Population: Participants analyzed consisted of subjects from the ITT cohort, defined as all subjects who were exposed to investigational product therapy and who provided baseline "sleep time" hot flash information and "sleep time" hot flash data for at least one post-baseline visit. Not all study subjects completed all data elements in their study diaries.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | 0.3 mg SCE-B Daily | 0.625 mg SCE-B Daily | Placebo Daily
Number analyzed (Participants) | 52 | 49 | 51
scores on a scale | 0.54 (0.066) | 0.56 (0.068) | 0.47 (0.067)

3. Secondary Outcome: Mean Change in Stanford Sleepiness Scale
Description: Change= Week 12 score - Baseline Score. Daytime sleepiness was derived from the subject self-assessment how they felt at a particular time of day. Subjects rated daytime sleepiness on the 7 point Stanford Sleepiness Scale (1=most alert to 7=sleepiest).
Time Frame: Baseline to End of Treatment (Week 12)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on Scale
Arm/Group | 0.3 mg SCE-B Daily | 0.625 mg SCE-B Daily | Placebo Daily
Number analyzed (Participants) | 47 | 49 | 48
Score on Scale | -0.79 (0.117) | -0.44 (0.117) | -0.62 (0.123)

4. Secondary Outcome: Mean Change in Biochemical Markers of Bone Metabolism (N-telopeptide).
Description: Change= Week 12 biochemical markers of bone metabolism (N-telopeptide) - Baseline biochemical markers of bone metabolism values for the intent-to-treat cohort.
Time Frame: From baseline to End of Treatment (Week 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nM BCE
Arm/Group | 0.3 mg SCE-B Daily | 0.625 mg SCE-B Daily | Placebo Daily
Number analyzed (Participants) | 45 | 41 | 42
nM BCE | -1.1 (6.67) | -3.8 (5.37) | -0.6 (7.53)

5. Secondary Outcome: Mean Change in Biochemical Markers of Bone Metabolism (Osteocalcin)
Description: Change= Week 12 biochemical markers of bone metabolism (Osteocalcin) - Baseline biochemical markers of bone metabolism values for the intent-to-treat cohort.
Time Frame: Baseline to End of Treatment (Week 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*ml
Arm/Group | 0.3 mg SCE-B Daily | 0.625 mg SCE-B Daily | Placebo Daily
Number analyzed (Participants) | 45 | 40 | 42
ng*ml | -3.7 (7.29) | -4.4 (7.94) | -0.3 (6.47)

6. Secondary Outcome: Mean Change in Biochemical Markers of Bone Metabolism (Sex Hormone Binding Globulin).
Description: Change= Week 12 biochemical markers of bone metabolism (Sex Hormone Binding Globulin) - Baseline biochemical markers of bone metabolism values for the intent-to-treat cohort.
Time Frame: Baseline to End of Treatment (12 weeks)
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: nmol/L
Arm/Group | 0.3 mg SCE-B Daily | 0.625 mg SCE-B Daily | Placebo Daily
Number analyzed (Participants) | 45 | 41 | 42
nmol/L | 19.5 (21.05) | 44.8 (38.86) | -3.3 (13.68)

ADVERSE EVENTS:
Time Frame: Adverse event reporting began on the first day of signing the informed consent and ended at the end of study drug treatment (approximately 16 weeks).
Description: Adverse events were reported during the subject's regularly scheduled visits at the investigational site.
Arm/Group | 0.3 mg SCE-B Daily | 0.625 mg SCE-B Daily | Placebo Daily
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/52 | 1/52
Other Adverse Events (participants affected / at risk) | 0/53 | 4/52 | 1/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.3 mg SCE-B Daily (N=53) | 0.625 mg SCE-B Daily (N=52) | Placebo Daily (N=52)
Right tibia and fibula shaft fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.3 mg SCE-B Daily (N=53) | 0.625 mg SCE-B Daily (N=52) | Placebo Daily (N=52)
Naspoharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can (i) review results communications prior to public release and can embargo communications regarding trial results for a period of at least 60 days but no more than 180 days from the time submitted to the sponsor for review; and (ii) require in instances of a multi-center study, that a single PI not disclose study data until after the multi-center results are published, provided such results are published within eighteen (18) months of the conclusion of the study.